CLINICAL TRIAL: NCT02247687
Title: Management of Participants With Low-level Persistent Viremia (ANRS 161 L-VIR)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment of participants for the study
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 161 L-Vir; 2014-001663-13 (EudraCT Number)
Record Dates: First submitted 2014-09-09; First posted 2014-09-25 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: HIV-1 Infection; Treatment Resistant Disorders; Viremia
Keywords: HIV-1; antiretroviral treatment; viral load
MeSH Terms: conditions — Viremia | interventions — Protease Inhibitors; Darunavir; Ritonavir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Counseling arm (Other): Counseling without antiretroviral treatment modification
  Interventions: Other: Counseling arm
- Switch arm for protease inhibitor (Active Comparator): Switch arm for protease inhibitor : intervention is the switch of current boosted protease inhibitor for Prezista® (darunavir)/ Norvir® (ritonavir) (switch for a drug with a higher genetic barrier) 600/100 mg two times a day (BID) with counseling.
  Interventions: Drug: Protease inhibitor
- Addition of Isentress® (raltegravir) (Active Comparator): Drug: Addition of Isentress® (raltegravir) arm
  • Addition of Isentress® (raltegravir) arm :Isentress® (raltegravir) 400 mg two times a day (BID) added to current antiretroviral treatment with counseling
  Interventions: Drug: Isentress® (raltegravir)

INTERVENTIONS:
Drug: Protease inhibitor — Modification in the antiretroviral treatment
  •Switch arm for protease inhibitor : intervention switch of current boosted protease inhibitor for Prezista® (darunavir)/ Norvir® (ritonavir) (switch for a drug with a higher genetic barrier) 600/100 mg two times a day (BID) with counseling.
  Other Names: Prezista® / Norvir®
  Arms: Switch arm for protease inhibitor
Drug: Isentress® (raltegravir) — • Addition of Isentress® (raltegravir) arm :Isentress® (raltegravir) 400 mg two times a day (BID) added to current antiretroviral treatment with counseling
  Arms: Addition of Isentress® (raltegravir)
Other: Counseling arm — No change of antiretroviral treatment but only counseling
  Arms: Counseling arm

SUMMARY:
Management of participants with low-level persistent viremia

DETAILED DESCRIPTION:
ANRS 161 L-Vir is a phase III prospective, randomized, multicenter, open-label, superiority trial for participants with low-level persistent viremia.

Participants will be randomized with a 1:1:1 ratio to the following three arms,

* Reference arm : counseling without antiretroviral treatment modification
* Switch arm : switch of current PI/r for Prezista® (darunavir)/ Norvir® (ritonavir) (switch for a drug with a higher genetic barrier) 600/100 mg two times a day (BID) with counseling.
* Addition of Isentress® (raltégravir) arm : Isentress® (raltegravir) 400 mg two times a day (BID) added to current antiretroviral treatment with counseling

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HIV-1 infection
* On combined antiretroviral regimen for at least 18 months
* Participant with a stable antiretroviral regimen for at least 6 months, including 2 Reverse-transcriptase inhibitor (INTI) + 1 Boosted Protease Inhibitor IP/r ,
* participant with at least 2 consecutive viral load between 50 and 500 copies/milliliter over the last 9 months (with at least 2 months between the two measurements) quantified with the same commercial kit.
* 50 <or= VL < 500 copies/milliliter at screening visit quantified with the same commercial kit than previous one.
* Participant naïve to raltegravir (RAL)
* failure of amplification or successful realization of genotypic resistance test without evidence for resistance mutations against current treatment (3TC/FTC accepted with M184V mutation)
* creatinin < 3 Upper Limit normal (ULN)
* Aspartate Amino Transférase (ASAT), Alanine Amino Transférase (ALAT) < 5 Upper Limit normal (ULN)
* hemoglobin > 8 g/dL
* platelets > 50 000/mm3
* In women, lack of current pregnancy verified by Beta Human Chorionic Gonadotropin (βHCG) at week -4 visit and use of a mechanical contraceptive method
* Informed consent
* Participants with an active health insurance coverage (article L1121-11 du Code de la Santé Publique)

Exclusion Criteria:

* HIV-2 infection,
* severe medical condition in the last month (inclusion is possible for a stable condition at screening)
* breastfeeding women, current pregnancy or planned pregnancy within 12 months.
* participant currently receiving Prezista® (darunavir)/ Norvir® (ritonavir) (600/100 mg) two times a day (BID) (of note, participants receiving Prezista® (darunavir)/ Norvir® (ritonavir) one time a day (QD) can be included)
* Hypersensitivity Prezista® (darunavir)/ Norvir® (ritonavir) or to any of the excipients of the study treatment
* participant under judicial protection (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship
* planned absence that could prevent the patient from participating in the trial (travel abroad, moving, pending work transfer ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in Virologic success by week 12 | week 12
  A virologic success is defined by a patient having plasma HIV-1 RNA levels <50 copies/ml at weeks 8 and 12.

SECONDARY OUTCOMES:
Proportion of participants with HIV-1 RNA < 50 copies/ml | week 4, week 8, week 12, week 24, week 36, week 48
Proportion of participants with HIV-1 RNA < 20 copies/ml | week 4, week 8, week 12, week 24, week 36, week 48
Proportion of participants with HIV-1 RNA <1copy/ml | week 8, week 12, week 24, week 36, week 48
Change in CD4 cells count from baseline | week 12, week 24, week 48 and end visit
  •Change was calculated as the CD4 count at the corresponding week minus the baseline CD4 count
Number of Participants With Virologic Failure and Emergence of Resistance | day 0 and visit at failure time
  •resistance patterns at failure time compared with day 0, in HIV-DNA and in HIV-RNA
Quantification of HIV DNA in peripheral blood mononucleated cell (PBMC) | day 0
  Quantification of HIV DNA in PBMC at day 0 and its association with the proportion of success in each arm
Levels of antiretroviral drugs in plasma | day 0 and end visit
  •plasma concentrations of antiretroviral drugs and correlation with success or failure of the strategy
Levels of antiretroviral drugs in hair | day 0, week 12, week 24and end visit
  •measurement of concentrations of antiretroviral drugs treatments in hair
Levels of HIV-1 RNA in seminal plasma | day 0, week 12, week 48 and end visit
  quantification of HIV RNA in seminal plasma
Incidence of Study interruption | From day 0 to week 24
  •proportion of participants who discontinued the strategy assigned by randomization at day 0 because of failure
Incidence of clinical and biological adverse events | from day 0 to week 48
  • proportions of participants experiencing a clinical or biological adverse events (ANRS scale)
Self-reported adherence | day 0, week 4, week 8, week 12, week 24, week 36, week 48 and end visit
  •self-reported percentage of antiretroviral treatment participant had taken during the last 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jade Ghosn, MD, PhD, Principal Investigator — APHP
Locations (20):
- France (20):
  - Hôpital Avicenne, Bobigny
  - Hôpital Jean Verdier, Bondy
  - Hôpital Saint André, Bordeaux
  - Hôpital Pellegrin, Bordeaux
  - Hôpital de la côte de Nacre, Caen
  - Hôpital Henry Mondor, Créteil
  - Hôpital Européen Georges Pompidou, France
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de l'Hôtel Dieu, Nantes
  - Hôpital Necker, Paris
  - Hôpital Tenon, Paris
  - Hôpital Hôtel Dieu, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital pitié Salpetrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Bichat, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicoll, Rouen
  - Hôpital Purpan, Toulouse